CLINICAL TRIAL: NCT03440099
Title: Sex-specific Adaptation to Different Resistance Exercise Programs in Older Adults
Brief Title: Sex-specific Adaptation to Resistance Training in Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Massachusetts, Amherst (Other)
Collaborators: University of Vermont (Other); National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 116-1974; 1R01AG047245-01A1 (NIH)
Record Dates: First submitted 2018-01-12; First posted 2018-02-20 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-05

CONDITIONS: Biological Aging
Keywords: Resistance Training; Sex Differences
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training (Other): All participants will participate in the 16-week resistance exercise training program.
  Interventions: Other: Resistance exercise training

INTERVENTIONS:
Other: Resistance exercise training — 16-week exercise training program, wherein one leg undergoes traditional low-velocity, high-load resistance training and the other leg undergoes high-velocity, low-load power training.

SUMMARY:
In general, men and women experience differing degrees of age-related decreases in physical function, with women having a greater prevalence of functional limitations and disability. A key predictor of this decrease in functional capacity is the reduction in leg muscle maximal power (product of force and velocity), which can be improved with exercise training. However, the development of exercise interventions to optimally improve skeletal muscle function in older adults has been difficult, in part because we now know that men and women respond differently to the same exercise training stimulus. In fact, the fundamental mechanisms by which habitual exercise improves physical function in older adults are still not well understood. The proposed studies are designed to address these knowledge gaps by examining the molecular and cellular mechanisms underlying the response to two distinct exercise training paradigms, and determining how these responses differ between older men and women. The investigators hypothesize that molecular, cellular and whole muscle contractile performance will be most improved in men by traditional low-velocity, high-load resistance training, and in women by high-velocity, low-load power training. Moreover, sex-specific structural responses in myofilament remodeling, protein expression and post-translational modifications will explain these sex-specific performance adaptations to each modality. To test these hypotheses, data will be gathered from 50 healthy, sedentary older men and women (65-75 years) prior to and following a 16-week unilateral exercise training program in which one leg undergoes resistance training and the other power training. The Specific Aims of this project are to identify the sex-specific effects of low-velocity resistance training versus high-velocity power training on: Aim 1) skeletal muscle function at the molecular, cellular and whole muscle levels, and Aim 2) protein expression and modification as well as size at the molecular and cellular levels. The within subject, unilateral intervention design provides a powerful model to minimize the effects of between-subject variability, and the translational approach will take advantage of our unique expertise with state-of-the-art measures from the molecular to whole body levels.

ELIGIBILITY:
Inclusion Criteria:

* Older adult (65-75 years old) volunteers will be healthy, by self-report, and sedentary, defined as no formal exercise program for the year prior to evaluation and < 2 sessions (30 min or more) of volitional exercise per week. Volunteers will be ambulatory without the use of walking aids and living independently in the community. All participants will be required to obtain a physician's consent to participate in the study, due to the exercise component, as is common practice in the Department of Kinesiology.

Exclusion Criteria:

* History of major neurological or neuromuscular condition that may impact physical function, including cerebrovascular disease, peripheral neuropathy, neurodegenerative disease, demyelinating disease, cerebellar or extrapyramidal disease, etc.
* History of myocardial infarction, angina, peripheral vascular disease, surgical or percutaneous coronary artery revascularization
* History of severe pulmonary disease (i.e., dyspnea that limits activities of daily living such as household ambulation and self-care)
* History of rheumatoid arthritis
* History of diabetes or other metabolic disease that may impact neuromuscular function
* Uncontrolled hypertension (blood pressure > 140/90)
* History of smoking in the past 1 year
* Moderate to severe lower extremity arthritis or pain (i.e., pain on level walking or that limits activities of daily living such as household ambulation and self-care)
* Pain, muscle cramps, joint stiffness, dyspnea, angina, light-headedness or other symptoms upon exertion
* The use of beta-blockers, sedatives, tranquilizers, or other medication that may impair physical function
* Individuals taking statin medications who report symptoms of muscle pain or myopathy
* Body-mass index >30 kg·m-2, as increased fat mass may alter single muscle fiber performance (Choi et al. J Gerontol A Biol Sci Med Sci 71:557-564, 2016)
* Body-mass index <18 kg·m-2, as this may be an early sign of frailty
* Must pass the Physical Activity Readiness Questionnaire for Everyone (PAR-Q+, in Appendix)
* Any persons taking anti-coagulant medication or with known coagulapathies will be excluded, due to increased bleeding risk from biopsy procedure
* Participants with a contraindication for magnetic resonance testing, including a pace-maker or other implant
* Women will be postmenopausal, as defined as cessation of menses for at least 12 months prior to study
* Men and women undergoing hormone replacement therapy, because this treatment may circumvent normal age-related declines in sex hormone levels (if taken hormone therapy must have been > 5 years ago)
* Unintentional weight loss of greater than 2.5 kg during the last 3 months
* Currently participating in or have participated in a weight loss or exercise training program in the last year
* An inability to understand written and spoken English
* An inability to follow instructions, as determined by the investigators during the consenting process

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in peak isokinetic power | This measure will be collected for each volunteer pre- and post-16 week exercise intervention and take approximately 30 minutes to collect for each time point.
  Peak isokinetic power at the whole muscle level will be evaluated using a dynamometer.
Change in single fiber specific power | This measure will be preformed on tissue biopsied from each volunteer pre- and post-16 week exercise intervention and requires approximately 1 week to collect per time point.
  Single fiber specific power will be measured from segments of chemically-skinned single human skeletal muscle fibers under maximal calcium-activated conditions, with muscle fiber type determined post-measurement by gel electrophoresis
Change in myosin attachment time | This measure will be preformed on tissue biopsied from each volunteer pre- and post-16 week exercise intervention and requires approximately one week to collect per time point.
  Myosin attachment time will be measured from segments of chemically-skinned single human skeletal muscle fibers under maximal calcium-activated conditions, with muscle fiber type determined post-measurement by gel electrophoresis.

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Miller, PhD, Principal Investigator — University of Massachusetts, Amherst
Locations (1):
- University of Massachusetts, Amherst, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Raw data will be considered for sharing under the rules indicated below. Raw datasets to be released for sharing will not contain identifiers. Data and associated documentation will be made available to users only under a signed and properly executed data-sharing agreement that provides for specific criteria under which the data will be used, including but not limited to a commitment to: 1) using the data only for research purposes; 2) securing the data using appropriate computer technology; and 3) destroying or returning the data after analyses are completed.
Time Frame: Research data will be made available upon final acceptance for publication of the major findings from the proposed studies.
Access Criteria: Data and associated documentation will be made available to users only under a signed and properly executed data-sharing agreement that provides for specific criteria under which the data will be used, including but not limited to a commitment to: 1) using the data only for research purposes; 2) securing the data using appropriate computer technology; and 3) destroying or returning the data after analyses are completed.

DOCUMENTS (3):
  • Study Protocol (2019-04-22): https://cdn.clinicaltrials.gov/large-docs/99/NCT03440099/Prot_004.pdf
  • Statistical Analysis Plan (2019-04-22): https://cdn.clinicaltrials.gov/large-docs/99/NCT03440099/SAP_005.pdf
  • Informed Consent Form (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT03440099/ICF_006.pdf